CLINICAL TRIAL: NCT00870831
Title: Islet Function and Clinical Analyses if Transplant Recipients (Project 2 of JDFI Washington University Center For Islet Transplantation) (Please Note That the JDRFI Funded Has Ended
Brief Title: Islet Function and Clinical Analyses of Transplant Recipients
Acronym: Islet OGTT
Status: Terminated | Type: Observational
Why Stopped: PI left University
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 00-0870
Record Dates: First submitted 2009-03-26; First posted 2009-03-27 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Type One Diabetes Mellitus
Keywords: diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples Without DNA — Serum samples are obtained during the OGTT and stored in a -20degree freezer. They are tested for Insulin C-peptide and glucose.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Islet Recipient: Subjects that have successfully received and maintained an Islet transplant at Washington University Center for Islet Transplantation
  Interventions: Other: OGTT (Oral Glucose Tolerance Test)
- Control: subjects that were similar in height, weight and age that did NOT have diabetes to act as the comparative group
  Interventions: Other: OGTT (Oral Glucose Tolerance Test)

INTERVENTIONS:
Other: OGTT (Oral Glucose Tolerance Test) — Subjects would consume 75grams of sugar (Dextrose, 10 oz) and blood samples taken at specified time points to measure glucose, insulin and C-peptide

SUMMARY:
To follow the patterns and natural history of Islet Transplant recipients (the ones that were involved in the Modified Edmonton Protocol) using oral glucose to check sugar levels as well as insulin and C-peptide over the course of 5 years

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes with hypoglycemia unawareness that received a Islet Transplant here at Washington University
* "control" subjects were matched to the transplant recipients base upon age, height, weight, & race (and could not have diabetes)

Exclusion Criteria:

* well controlled Type 1 diabetes
* transplant failure
* unable to match potential subject to a recipient

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Type 1 diabetics that have successfully received and maintained an islet transplant here at Washington University. Loss of transplant function is an exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2000-10; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
OGTT will be performed every 6 months for 5 years in subjects with a functioning Islet Transplant | 5 years

SECONDARY OUTCOMES:
The OGTT reflects the function of the Islet transplant and could be used as an indication of Islet Transplant function | 5yrs

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth S Polonsky, MD, Principal Investigator — Washington University School of Medicine; Daniel C Brennan, MD, Principal Investigator — Washington University School of Medicine